CLINICAL TRIAL: NCT04286126
Title: Individualized Neuroimaging Biomarkers for Predicting rTMS Response in OCD
Brief Title: Neuroimaging Biomarkers for Predicting rTMS Response in OCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Ian Kratter, Clinical Assistant Professor, Department of Psychiatry & Behavioral Sciences, Stanford University School of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53879
Record Dates: First submitted 2020-02-21; First posted 2020-02-26 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: transcranial magnetic stimulation; theta burst
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- bilateral DMPFC (Active Comparator): This arm will receive intermittent theta-burst stimulation to bilateral DMPFC site.
  Interventions: Device: Active bilateral DMPFC
- right OFC (Active Comparator): This arm will receive continuous theta-burst stimulation to the right OFC site.
  Interventions: Device: Active right-sided OFC

INTERVENTIONS:
Device: Active bilateral DMPFC — Participants in this arm will receive rTMS to bilateral DMPFC. The DMPFC will be targeted utilizing either Nexstim's eField neuronavigation system or Localite's neuronavigation system. Stimulation intensity will be standardized at 100% of resting motor threshold (RMT).
  Arms: bilateral DMPFC
Device: Active right-sided OFC — Participants in this arm will receive rTMS to the right OFC. The right OFC will be targeted utilizing either Nexstim's eField neuronavigation system or Localite's neuronavigation system. Stimulation intensity will be standardized at 110% of resting motor threshold (RMT).
  Arms: right OFC

SUMMARY:
This study evaluates an accelerated schedule of theta-burst stimulation using a Transcranial Magnetic Stimulation (TMS) device for treatment-resistant Obsessive Compulsive Disorder (OCD). In a randomized fashion, half the participants will receive accelerated theta-burst stimulation at the dorsomedial prefrontal cortex (DMPFC), while half will receive accelerated theta-burst stimulation at the right orbitofrontal (rOFC) site.

DETAILED DESCRIPTION:
Medications (SSRIs and D2 antagonists) and cognitive-behavioral therapy are the mainstays of treating OCD; however, many patients show only a partial response, and more than 25% of patients show no improvement with these treatments. Repetitive transcranial magnetic stimulation (rTMS) is a promising alternative, using powerful, focused magnetic field pulses to stimulate target brain areas. So far, at least two stimulation targets have consistent evidence of efficacy in OCD: the dorsomedial prefrontal cortex (DMPFC) and the orbitofrontal cortex (OFC). Patients often show a strong response to one target but not the other. It is not well understood why some patients respond, while others do not.

The investigators previously developed methods for discovering neurophysiological subtypes of depression based on resting state functional Magnetic Resonance Imaging (fMRI) measures of functional connectivity (RSFC) in relevant brain networks; diagnosing them in individual patients; and using them to predict individual differences in rTMS response. Subsequently, motivated by recent studies characterizing individual variability in the topology of these functional networks, the investigators have optimized methods for improving the accuracy of these predictions by accounting for individual variability, stabilizing the selection of treatment-predictive features, and increasing robustness in replication samples through regularization. Here, the investigators propose applying these methods to discover novel network-based subtypes of OCD and develop prognostic neuroimaging biomarkers for predicting differential treatment response to rTMS targeting the DMPFC or OFC, which could subsequently be tested in a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. meets Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for OCD with a moderate level of severity as defined by a Yale-Brown Obsessive Compulsive Scale (YBOCS) score of at least 18.
2. stable on Serotonin Re-uptake Inhibitor (SRI) medication for at least 8 weeks prior to (with plans to continue throughout) the study Note: Medications that are known to increase cortical excitability (e.g., buprorion, maprotiline, tricyclic antidepressants, classical antipsychotics) or to have an inhibitory effect on brain excitability (e.g., anti-convulsants, benzodiazepines, and atypical antipsychotics), or any other medications with relative hazard for use in TMS will be allowed upon review of medications and/or motor threshold determination by TMS specialist.
3. failed at least 1 prior trial of standard first-line OCD treatment per American Psychological Association (APA) Practice Guidelines (serotonin reuptake inhibitor [SRI] or cognitive behavioral therapy with exposure and response prevention)OR had refused these treatments for individual reasons.
4. capacity to provide informed consent.
5. ability to tolerate clinical study procedures.
6. successfully complete the screening forms at the Stanford Center for Cognitive and Neurobiological Imaging (CNI) without any contraindications.

Exclusion Criteria:

1. Current psychosis (re-assessed only if screening appointment was more than 30 days ago - Structured Clinical Interview for DSM-IV (SCID) - 5 Module B)
2. Current bipolar disorder (assessed during baseline if screening appointment was more than 30 days ago - SCID-5 Module D)
3. Severe depression [Note: 17-item Hamilton Depression Rating Scale (HDRS-17) must be less or equal to 20 to enter study, assessed during baseline if last assessment was more than 1 week ago]
4. Current active suicidality (as determined by C-SSRS at baseline of 3 or above)
5. Current moderate or severe Alcohol Usage Disorder or Substance Usage Disorder (except nicotine and caffeine) according to the DSM-5 criteria (assessed only if screening appointment was more than 12 months ago - SCID-5 Module E)
6. Current eating disorder (assessed during baseline if screening appointment was more than 3 months ago - SCID-5 Module I)
7. History of seizure, having an EEG, stroke, head injury (including neurosurgery), implanted devices, frequent or severe headaches, brain related conditions (e.g., intracranial mass lesions globe injuries, hydrocephalus), illness that caused brain injury or first degree relative with seizure disorder (assessed during screening via medical history assessment and TMS Safety Screen by study MD)
8. Individuals with primary hoarding disorder without a DSM-5 OCD diagnosis (as determined by SCID-5 and YBOCS checklist assessed only if screening appointment was more than 30 days ago)
9. Planning to commence Cognitive Behavioral Therapy (that includes exposure and response prevention) during the period of the study or have begun Cognitive Behavioral Therapy within 8 weeks prior to enrollment (assessed during baseline by study MD)
10. Pregnant or nursing females (assessed via urine dipstick if screening appointment was more than 30 days ago)
11. Positive urine screen for illicit drugs (assessed via urine dipstick if screening appointment was more than 30 days ago) [Exceptions: (1) any prescribed medication that participant is currently taking and (2) positive cocaine metabolite after consumption of coca tea]
12. History of any implanted device or psychosurgery (assessed during baseline by study MD)
13. History of receiving Electroconvulsive Therapy (ECT) (assessed during baseline by study MD)
14. Age of OCD symptom onset >30

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage change in Yale-Brown Obsessive-Compulsive Scale (YBOCS) | Baseline (Pretreatment) to immediate post-treatment follow up
  The YBOCS is a 10-item clinician-rated questionnaire that assesses the impact and severity of an individual's obsessive thoughts and compulsive behaviors. The minimum and maximum scores are 0 and 36, respectively, with higher score indicating greater severity.

SECONDARY OUTCOMES:
Percent change in the Obsessive-Compulsive Inventory-Revised (OCI-R) | Baseline (Pretreatment) to immediate post-treatment follow up
  The Obsessive-Compulsive Inventory-Revised (OCI-R) has 18 items. Each item can be scored on a 5 point scale from 0 to 4. Total score can range from 0 to 72, with higher scores indicating more severe OCD.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Kratter, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Department of Psychiatry and Behavioral Sciences, Stanford School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Chung SW, Hill AT, Rogasch NC, Hoy KE, Fitzgerald PB. Use of theta-burst stimulation in changing excitability of motor cortex: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2016 Apr;63:43-64. doi: 10.1016/j.neubiorev.2016.01.008. Epub 2016 Feb 3. PMID 26850210
- [Background] Jelic MB, Milanovic SD, Filipovic SR. Differential effects of facilitatory and inhibitory theta burst stimulation of the primary motor cortex on motor learning. Clin Neurophysiol. 2015 May;126(5):1016-23. doi: 10.1016/j.clinph.2014.09.003. Epub 2014 Sep 16. PMID 25281475
- [Background] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537
- [Background] Plewnia C, Pasqualetti P, Grosse S, Schlipf S, Wasserka B, Zwissler B, Fallgatter A. Treatment of major depression with bilateral theta burst stimulation: a randomized controlled pilot trial. J Affect Disord. 2014 Mar;156:219-23. doi: 10.1016/j.jad.2013.12.025. Epub 2013 Dec 28. PMID 24411682
- [Background] Prasser J, Schecklmann M, Poeppl TB, Frank E, Kreuzer PM, Hajak G, Rupprecht R, Landgrebe M, Langguth B. Bilateral prefrontal rTMS and theta burst TMS as an add-on treatment for depression: a randomized placebo controlled trial. World J Biol Psychiatry. 2015 Jan;16(1):57-65. doi: 10.3109/15622975.2014.964768. Epub 2014 Nov 28. PMID 25430687
- [Background] Daskalakis ZJ. Theta-burst transcranial magnetic stimulation in depression: when less may be more. Brain. 2014 Jul;137(Pt 7):1860-2. doi: 10.1093/brain/awu123. Epub 2014 May 15. No abstract available. PMID 24833712
- [Background] Thut G, Pascual-Leone A. A review of combined TMS-EEG studies to characterize lasting effects of repetitive TMS and assess their usefulness in cognitive and clinical neuroscience. Brain Topogr. 2010 Jan;22(4):219-32. doi: 10.1007/s10548-009-0115-4. Epub 2009 Oct 28. PMID 19862614
- [Background] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360
- [Background] Fung PK, Robinson PA. Neural field theory of synaptic metaplasticity with applications to theta burst stimulation. J Theor Biol. 2014 Jan 7;340:164-76. doi: 10.1016/j.jtbi.2013.09.021. Epub 2013 Sep 21. PMID 24060620
- [Background] Biswal B, Yetkin FZ, Haughton VM, Hyde JS. Functional connectivity in the motor cortex of resting human brain using echo-planar MRI. Magn Reson Med. 1995 Oct;34(4):537-41. doi: 10.1002/mrm.1910340409. PMID 8524021
- [Background] Greicius MD, Krasnow B, Reiss AL, Menon V. Functional connectivity in the resting brain: a network analysis of the default mode hypothesis. Proc Natl Acad Sci U S A. 2003 Jan 7;100(1):253-8. doi: 10.1073/pnas.0135058100. Epub 2002 Dec 27. PMID 12506194
- [Background] Fox MD, Snyder AZ, Vincent JL, Corbetta M, Van Essen DC, Raichle ME. The human brain is intrinsically organized into dynamic, anticorrelated functional networks. Proc Natl Acad Sci U S A. 2005 Jul 5;102(27):9673-8. doi: 10.1073/pnas.0504136102. Epub 2005 Jun 23. PMID 15976020
- [Background] Greicius MD, Supekar K, Menon V, Dougherty RF. Resting-state functional connectivity reflects structural connectivity in the default mode network. Cereb Cortex. 2009 Jan;19(1):72-8. doi: 10.1093/cercor/bhn059. Epub 2008 Apr 9. PMID 18403396